CLINICAL TRIAL: NCT07070804
Title: Maternal Biomarkers and Environmental Contributors to Autism Spectrum Disorders in Children of First-time Mothers
Status: Not yet recruiting | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, David Haas, Professor of Medicine, Indiana University
Other Study IDs: nuMoM2bAutism
Record Dates: First submitted 2025-06-27; First posted 2025-07-17 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Autism
Keywords: nuMoM2b; autism; prediction
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — urine for future use
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: None-placebo — No interventions performed

SUMMARY:
This study will recruit nuMoM2b participants to complete autism screening surveys and will identify 200 children with autism and 400 controls for the study. It will then use existing biospecimens to measure pesticides in maternal urine and metabolomic urine and cord blood predictors of autism risk. All data will then be used to build a predictive model for autism risk at the child's birth.

DETAILED DESCRIPTION:
NuMoM2b participans will be contacted as part of ongoing contacts and will be consented for their offspring to participate. The children will also undergo an Assent process. Screening for autism will occur using standard validated tools and anyone who screens positive will have remote diagnostic testing with trained study staff. The study aims to identify a cohort of 200 children with autism and will then randomly select a group of 400 children typically developing. Predictive models for autism will be constructed using pregnancy and birth data as well as biomarkers from maternal urine and cord blood. We will include metabolomic biomarkers as well as environmental exposures to assess if they improve the predictive model.

ELIGIBILITY:
Inclusion Criteria:

* child of nuMoM2b study participant

Exclusion Criteria:

* no biological samples collected during pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: children of nuMoM2b cohort
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2028-08-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of autims | The children are age 11-14 currently. The outcome will be measured during contact with the children in the first 18 months of the project.
  Autism diagnoses will be made using the Autism Diagnostic Inventory on all children who screen positive. Alternatively, if already diagnosed clinically, we will request the diagnostic tool used previously for the child.

IPD SHARING:
Plan to Share IPD: Yes
deidentified data upon request per NIH guidance
Supporting Information: Study Protocol
Time Frame: After study completion